CLINICAL TRIAL: NCT06122038
Title: Impact of Powdered Tart Cherries on Recovery From Repeated Sprints in Trained Males and Females
Brief Title: Impact of Powdered Tart Cherries on Recovery From Repeated Sprints
Acronym: TCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-23-11
Record Dates: First submitted 2023-05-15; First posted 2023-11-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2024-04

CONDITIONS: Inflammation; Oxidative Stress; Soreness, Muscle; Muscle Damage
Keywords: Tart Cherry; Inflammation; Muscle Soreness; Muscle Damage
MeSH Terms: conditions — Inflammation; Myalgia

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized, double-blind, placebo group study design
Who Masked: Participant, Investigator
Masking Description: In a double-blind, placebo-controlled fashion, participants will be randomly assigned to one of two supplementation groups. One group will be assigned to ingest rice flour which will serve as a placebo group. The other group will be assigned to ingest 500 mg/day of Tart Cherry Extract Powder (ADSO Naturals). All study materials will be prepared into gelatin capsules of identical size, color, shape, and transparency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Rice Flour. Dispensed during visit 1. Participants will consume 1 dose per day for 10 days.
  Interventions: Dietary Supplement: Placebo
- Tart Cherry Extract Powder (Experimental): Tart Cherry Extract Powder (ADSO Naturals). Dispensed during visit 1. Participants will consume 1 dose per day for 10 days.
  Interventions: Dietary Supplement: Tart Cherry Extract Powder

INTERVENTIONS:
Dietary Supplement: Tart Cherry Extract Powder — Tart Cherry Extract Powder (ADSO Naturals). Dispensed during visit 1. Participants will consume 1 dose per day for 10 days.
  Arms: Tart Cherry Extract Powder
Dietary Supplement: Placebo — Rice power placebo. Dispensed during visit 1. Participants will consume 1 dose per day for 10 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate changes in force and power production, soreness, inflammation, and oxidative stress after repeated sprinting activity and powdered tart cherry ingestion in trained males and females.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate changes in force and power production, soreness, inflammation, and oxidative stress after repeated sprinting activity and powdered tart cherry ingestion in trained males and females. This study will utilize a randomized, double-blind, placebo group study design. Prior to any data collection, potential participants will be explained the protocol and then review and sign an IRB-approved consent form. Healthy male and female (n=40) participants who report regularly practicing or competing in high-intensity multi-modal resistance based exercise will complete the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (n=40) participants between the ages of 18 - 35 years of age will finish the study protocol. An even distribution of males (n=20) and females (n=20) is planned.
* Participating in some form of exercise at least four days per week with at least two days consisting of some form of high-intensity exercise for the past six months.
* Examples include regular gym attendance to complete resistance training, interval exercise, or participation in some form of organized physical activity involving high-speed running or other forms of high-intensity exercise.
* Have a body mass index (BMI) range of 18.0 - 30.0 kg/m2. Males with a body mass index greater than 30.0 kg/m2, but a body fat percentage less than 27.5% fat will be accepted into the study. Females with a body mass index greater than 30.0 kg/m2, but a body fat percentage less than 32.5% fat will be accepted into the study.

Exclusion Criteria:

* Participant has a positive medical history of heart disease/cardiovascular disease, uncontrolled hypertension (140/90 or greater mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease, or Type I or Type II diabetes.
* Participant has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within five years prior to screening visit.
* Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
* Positive medical history for any neurological condition or neurological disease
* Currently smoke or have quit within the past six months
* Current daily use of aspirin, NSAIDS, naproxen sodium, COX-2 inhibitors, or any other over-the-counter or prescribed medication indicated for pain relief.
* Intake of any dietary supplement known or purported to impact muscle repair and recovery such as antioxidants, curcumin, turmeric, branched-chain amino acids, vitamin D, tart cherry, pomegranate, fish oils, or creatine monohydrate.
* Individuals who indicate they are actively involved in any form of a dietary program in the past 30 days to lose weight
* Participants who are lactating, pregnant or planning to become pregnant
* Have a known sensitivity or allergy to any of the study products
* Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data
* History of alcohol or substance abuse in the 12 months prior to screening
* Receipt or use of an investigational product in another research study within 28 days prior to baseline testing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Counter movement Jump Height | 10 days
  Jump height from counter movement jump
Counter movement jump peak propulsive force (N) | 10 days
  Peak propulsive force (N) from counter movement jump
Counter movement jump relative breaking force (N) | 10 days
  relative breaking force (N/kg) from counter movement jump
Isokinetic knee extension maximal voluntary contraction. | 10 days
  Peak isokinetic knee extension force (N) from a isokinetic knee extension exercise using a Biodex System 3
Isometric mid-thigh pull maximal voluntary contraction | 10 days
  Isometric maximal voluntary contraction peak force will be measured using an isometric mid-thigh pull assessment. Peak force production will be measured in Newtons.
Perceived recovery Visual Analog Scale | 10 days
  Perceived recovery Visual Analog Scale ranging from 0 (worst) to 100 (best)
Perceived soreness Visual Analog Scale | 10 days
  Perceived soreness Visual Analog Scale ranging from 0 (worst) to 100 (best)
Pain to Pressure threshold | 10 days
  Pain to Pressure threshold from algometry (higher = less sore). Minimum values are 0 N, maximum values are 110 N
Changes in Creatine Kinase concentrations | 10 days
  Changes in Creatine kinase concentrations following damaging exercise
Changes in Creatine Kinase-myocardial band concentrations | 10 days
  Changes in Creatine kinase-myocardial band concentrations following damaging exercise
Sprint time | Baseline
  Fastest and average sprint time during 15 30-meter sprint recorded using digitally timed timing gates

SECONDARY OUTCOMES:
Peak power | 10 days
  Peak power during a wingate anaerobic test
Changes in Protein carbonyls concentration | 10 days
  Protein carbonyls concentration changes
Changes in 8-isoprostane concentration | 10 days
  8-isoprostane concentration changes
Changes in testosterone-cortisol ratio | 10 days
  Testosterone-cortisol ratio changes
Changes in TNF-alpha concentration | 10 days
  Changes in TNF-alpha concentration
Changes in IL-6 concentration | 10 days
  Changes in IL-6 concentration
Changes in IL-10 concentration | 10 days
  Changes in IL-10 concentration
Desire to exercise visual analog scale | 10 days
  Desire to exercise visual analog scale (0 = not ready to train, 100 = very ready to train)
Pittsburgh sleepiness Scale Score | 10 days
  Pittsburgh sleepiness Scale Score (lower scores indicate higher level of sleepiness)
Changes in Uric Acid Concentrations | 10 days
  Changes in Uric Acid concentrations

OTHER OUTCOMES:
Resting Heart Rate | 10 days
  Resting heart rate at all study visits
Resting Blood pressure | 10 days
  Resting Blood pressure at all study visits
Reported Adverse Events | 10 days
  Self-Reported Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No